CLINICAL TRIAL: NCT04139850
Title: The Establishment of Korean Hepatitis B Patients Cohort
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0748
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; cohort; nationwide; prospective; antiviral therapy
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — 16cc of whole blood sample in CPT tube
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Korean chronic hepatitis B patients cohort: Korean patients with chronic hepatitis B with or without antiviral therapy on a regular follow-up in tertially medical institution
  Interventions: Drug: Discontinuation of antiviral treatment in chronic hepatitis B cohort patients

INTERVENTIONS:
Drug: Discontinuation of antiviral treatment in chronic hepatitis B cohort patients — For the selective patients in the cohort with long-term antiviral therapy and with conditions such as HBeAg negative or loss more than one year, antiviral therapy is able to be discontinued with an intensive inspection who agreed to the process. If there are need of this intervention, another multicenter IRB approval will be taken.

SUMMARY:
According to the World Health Organization about 1,400,000 deaths reported annually, are related to chronic liver disease. Chronic liver disease is very prevalent in South Korea, placing a large economic burden nationwide. Subsequently, an effective and systematized approach to managing chronic hepatitis is imperative in Korea.

The natural history of chronic liver disease differs greatly according to race and ethnicity. However, there is scarcity of epidemic data on chronic hepatitis based on Korean patients. Therefore, the investigators plan to establish a prospective multicenter cohort for chronic hepatitis B based on Korean patients that may be utilized for various future clinical studies on chronic hepatitis B in Korea, and thereby serve as a basis for the establishment and distribution of clinical guidelines for Korean patients with chronic hepatitis B, as part of a nationwide project supported by the Centers for Disease Control (CDC), Korea.

The investigators plan to collect more than 2,000 cases per year with 6 months of regular follow-up interval as have been advised by the CDC during 10 years of the study period (from Sep. 2015) from 5 tertiary hospitals located in Korea. The investigators plan to register available cases from those who are available to agree to give written informed consent and provide their blood samples to participate in this study prospectively, according to the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. age above 19 years;
2. CHB diagnosis with more than 6 months of HBsAg positive;
3. Patients who followed up regularly by medical institutions due to CHB;
4. Patients who can be followed up according to the research protocol;
5. Patients who have consented to the written consent of the applicant or guardian.

Exclusion Criteria:

1. HCC diagnosis before enrollment;
2. Malignant tumor other than HCC within 5 years;
3. Hepatitis C virus or human immunodeficiency virus co-infection;
4. Fatal conditions such as decompensated liver function, end stage renal disease and severe heart failure;
5. not be suitable for the research purpose.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic in tertiary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-09-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Development of liver cirrhosis, decompensation or liver cancer | Time of registration of patient to cohort complement (10 years)
  This study aims for the establishment of chronic hepatitis B cohort and has no other primary end point other than the registration of the patient. (For Time-to-Event outcome measures, the development of events including HCC, ascitic decompensation, variceal bleeding, hepatic encephalopathy, transplantation, and death will be followed up to 10 years after enrollment. Time to the development of each kind of event will be calculated from the date of enrollment and the respective date of event development.) Safety issue: No

SECONDARY OUTCOMES:
Safety and efficacy for patients with or without antiviral therapy | Time of registration of patient to cohort complement (10 years)
  Virologic response, HBsAg loss or seroconversion, development of resistance to medication, side effect with or without antiviral therapy Virologic breakthrough/development of liver cirrhosis, decompensation or HCC after discontinuation of antiviral therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The patients' clinical and laboratory information are stored in the Korean CDC database as a form of eCRF, then be locked after data cleaning. The sharing data will be coded and won't include patients' sensitive individual information such as a unit-ID and name. The coded data and saved samples will be provided for the guaranteed researchers by the government after confirmation of the relevance of their clinical and basic researches plan related with HBV, during the study and after the study ends.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code